CLINICAL TRIAL: NCT00220454
Title: Effect of Estrogen on the Stress Response for Postmenopausal Women
Brief Title: Effect of Estrogen & Stress for Postmenopausal Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seattle Institute for Biomedical and Clinical Research (Other)
Collaborators: National Alliance for Research on Schizophrenia and Depression (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RDIS 0007; Baker-Y02 (Sponsor); BL17 (Supporting Institution)
Record Dates: First submitted 2005-09-19; First posted 2005-09-22 (Estimated); Last update posted 2007-02-27 (Estimated); Status verified 2007-02

CONDITIONS: Aging
Keywords: cognition; estradiol; cortisol; postmenopause
MeSH Terms: interventions — Estradiol; Hydrocortisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Climara
Drug: Hydrocortone

SUMMARY:
The study tests the hypothesis that estradiol administration exacerbates the effects of the stress hormone cortisol on cognition and mood for postmenopausal women. This randomized, placebo-controlled, double-blind study was designed to examine the effects of an eight-week trial of transdermal estradiol replacement therapy (0.10 mg/day) in combination with 4 days of oral hydrocortisone (90 mg/day in 3 daily doses of 30 mg per dose) in the last week of hormone therapy on cognition and mood in healthy postmenopausal women. Forty cognitively healthy postmenopausal women were randomized to receive either placebo or estradiol skin patches for 8 weeks. In the middle of the 7th week (day 57), subjects in each group were again randomized to receive either a placebo tablet or an oral hydrocortisone tablet 3x/day for 4 days. Memory testing and blood collection occurred at baseline, at week 4, and again at week 8.

DETAILED DESCRIPTION:
Estrogen replacement has been associated with improved learning and memory in both animal and human studies. However, there is some evidence to suggest that "stress" has a detrimental effect on learning for female animals who still have naturally circulating estrogen. Interestingly, when the effects of this hormone are blocked in the body, stress no longer impairs learning. Several investigators have raised the possibility that the physiological response to stress may be exaggerated for women compared to men. Gender differences in biological systems that control the release of gonadal and stress hormones may explain why estrogen is beneficial for women under nonstressed conditions, but detrimental for them under stressed conditions. To date, no study has carefully controlled or manipulated both estrogen use and cortisol levels to further explore this issue. In this placebo-controlled, double blind, parallel-group design clinical study we will evaluate whether estrogen use exacerbates stress-related impairments in cognition for healthy postmenopausal women. Forty subjects will receive either 0.10 mg/day of transdermal beta-estradiol or a placebo skin patch for 8 weeks. In the last week of treatment, subjects will receive 90 mg/day of oral hydrocortisone or a placebo for 4 consecutive days. Scores on tests of memory, attention, and mood, as well as blood levels of estrogen and cortisol will be assessed at baseline, and at weeks 4 and 8. We predict that the estrogen+cortisol combination will have a deleterious effect on cognition and mood relative to the effects of either hormone administered alone. The results of this study are likely to provide important information regarding not only the nature of the interaction between these hormonal systems that occurs in response to stress, but also the conditions under which the beneficial effects of estrogen may be overshadowed.

ELIGIBILITY:
Inclusion Criteria:

Postmenopausal women

Exclusion Criteria:

Current HRT use Hx of DVT current steroid user Cushing's or other similar disease Breast or uterine cancer

Ages: 55 Years to 90 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2002-12; Study Completion 2005-03

PRIMARY OUTCOMES:
Change in cognitive test scores at months 1 & 3 vs. baseline

SECONDARY OUTCOMES:
Correlation between change in blood levels of cortisol & estradiol and cognitive scores
Correlation between change in cognitive score and treatment-induced change in beta-amyloid

CONTACTS AND LOCATIONS:
Overall Officials: Laura D Baker, PhD, Principal Investigator — VA Puget Sound Health Care System & University of Washington